CLINICAL TRIAL: NCT04546854
Title: Influenza 2020/2021. A Survey to Assess How People's Political Attitudes and Messages Influence Their Behavioral Intentions in the United Kingdom.
Brief Title: Influenza 2020/2021
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warwick (Other)
Responsible Party: Principal Investigator, Kelly Ann Schmidtke, Assistant Professor, University of Warwick
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BSREC 167/19-20
Record Dates: First submitted 2020-09-05; First posted 2020-09-14 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Influenza Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative - Binding Appeal (Experimental)
  Interventions: Behavioral: Appeals
- Liberal - Individulizing Appeal (Experimental)
  Interventions: Behavioral: Appeals

INTERVENTIONS:
Behavioral: Appeals — Written text motivating participants to take up the seasonal influenza vaccination

SUMMARY:
As part of the fight against COVID-19, the UK government has announced its most comprehensive flu campaign to date (https://www.gov.uk/government/news/most-comprehensive-flu-programme-in-uk-history-will-be-rolled-out-this-winter). This should not be surpising: every year NHS hospitals experience an overwhelming number of influenza cases, and COVID-19 increases this concern. As in previous years, the flu vaccine is free at the point of care for people 65 and over. New this year is that later in the season the vaccine will be made available free at the point of care for people 50 and over. However, if people refuse to take the vaccine this comprehensive program cannot benefit public health.

The degree to which vaccine hesitancy is expressed varies across characteristics of the vaccine considered and the time and place it is offered, and across characteristics of the person's perceptions of complacency, convenience, confidence, calculations, and communal responsibility, i.e. the "5Cs". Information campaigns can be used to influence all 5Cs, and public facing information is often a necessary component of public health campaigns that may also include structural components. Largely, information campaigns can be viewed as a type of educational intervention.

Educational interventions may fall short of what is needed to alter people's intentions to vaccinate where they focus on system 1 rational thinking processes and neglect system 2 automatic thinking processes. To be more effective, public health messages must be tailored to align with the "beliefs, attitudes, and motivations" of the very people they intend to influence.

Fact-led educational interventions to increase parents' intentions to vaccinate their children are particularly ineffective where more subtle content opposes the recipient's deep-seated values. In a different context, recycling behaviour, previous research demonstrated that messages aligned with people's deep-seated values (i.e. the moral foundations that underlie political ideologies) are more likely to promote desired behavioural intentions than unaligned messages.

The present research expands the scope of previous research in two ways. First, rather than investigating parental attitudes towards vaccination, the investigators will look at people's intentions to self-vaccinate. Second, the investigators will explore the effectiveness of messages aligned with the moral foundations that underlie individual's political ideologies on their intentions to be vaccinated.

ELIGIBILITY:
Inclusion Criteria:

* Resident in England
* Age 50+ years old, inclusive

The age criteria is set at 50+ years old, because this is the age group currently being advised by Public Health England to seek the flu jab as soon as possible this season. (https://www.gov.uk/government/news/most-comprehensive-flu-programme-in-uk-history-will-be-rolled-out-this-winter).

Exclusion Criteria:

* Not a resident in England
* Age less than 50 years old

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
Intentions to take up the seasonal influenza vaccination | 1 day
  Participants rate their intentions to take up the seasonal influenza vaccination on a 7-point likert scale, from strongly disagree (=1) to strongly agree (=7).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Warwick, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT04546854/Prot_000.pdf